CLINICAL TRIAL: NCT06052306
Title: A Phase 1 Open-label, First-in-human, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Actinium-225-macropa-pelgifatamab (BAY 3546828) in Participants With Advanced Metastatic Castration Resistant Prostate Cancer (mCRPC)
Brief Title: A Study to Learn How Safe the Study Treatment Actinium-225-macropa-pelgifatamab (BAY3546828) is, How it Affects the Body, How it Moves Into, Through and Out of the Body, and About Its Anticancer Activity in Participants With Advanced Metastatic Castration-resistant Prostate Cancer (mCRPC)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22143; 2022-502623-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-09-07; First posted 2023-09-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dose escalation of BAY3546828 (Experimental): Participants with advanced metastatic castration-resistant prostate cancer (mCRPC) will receive 225Ac-pelgi dose in a stepwise fashion, according to a predefined dose escalation scheme
  Interventions: Drug: BAY3546828
- Dose expansion group A of BAY3546828 (Experimental): Participants with advanced mCRPC with at least 1 but no more than 2 prior taxane regimens. No prior radionuclide therapy
  Interventions: Drug: BAY3546828
- Dose expansion group B of BAY3546828 (Experimental): Participants with advanced mCRPC who have not received taxane chemotherapy since becoming castration-resistant. No prior radionuclide therapy.
  Interventions: Drug: BAY3546828
- Dose expansion group C of BAY3546828 (Experimental): Participants with advanced mCRPC after prior Lutetium-177 labeled PSMA ligand (177Lu-PSMA) treatment.
  Interventions: Drug: BAY3546828

INTERVENTIONS:
Drug: BAY3546828 — Intravenous (IV) infusion on Day 1 of each cycle.

SUMMARY:
Researchers are looking for a better way to treat people who have advanced metastatic castration-resistant prostate cancer (mCRPC). In participants with metastatic castration-resistant prostate cancer (mCRPC), the cancer of the prostate has spread to other parts of the body (metastatic) and does not respond to the lowering of testosterone levels in the body (castration resistant). The cancer is 'advanced' and is unlikely to be cured or controlled with currently available treatments. Despite new treatment options for participant(s) with prostate cancer in recent years, the cancer often returns and worsens.

The study treatment actinium-225-macropa-pelgifatamab (also called 225Ac-pelgi or BAY3546828) is a new type of treatment under development for participants with mCRPC who have already received available treatments or have few treatment options available. It works by binding to a protein on the surface of the cancer cells called prostate specific membrane antigen (PSMA). As it gives off a type of radioactivity that travels a very short distance, it kills the nearby (cancer) cells that express PSMA.

The main purpose of this first-in-human study in participants with mCRPC is to learn:

* How safe different doses of 225Ac-pelgi are.
* To what degree medical problems caused by 225Ac-pelgi can be tolerated by the participants?
* Which dose of 225Ac-pelgi is optimal for treatment (safe and working well)?
* How good is 225Ac-pelgi's anticancer activity?

To answer this, the researchers will look at:

* The number and severity of medical problems that the participants have after treatment with 225Ac-pelgi (per dose level).
* The ratio of medical problems and anticancer activity per dose.
* Anticancer activity of the optimal 225Ac-pelgi dose as proportion of participants who have at least halved prostate-specific antigen (PSA) levels after 12 weeks of treatment or later and/or shrunken or no longer detectable tumors.
* The lowest PSA level reached after treatment start.

Doctors keep track of all medical problems (also called adverse events) that participants have during the study, even if they do not think that they might be related to the study treatment.

Anticancer activity is measured using cancer imaging techniques and change in blood level of a protein called PSA. PSA is made by normal and by cancerous cells in the body. The PSA level is taken as a marker for prostate cancer development and is usually elevated in participants with mCRPC.

In addition, researchers want to find out how 225Ac-pelgi moves into, through and out of the body.

The study will have two parts. The first part, called dose escalation, is done to find the most appropriate dose and schedule that can be given in the second part of the study. For this, each participant will receive one of the predefined increasing doses of 225Ac-pelgi as an infusion into the vein. All participants in part 2, called dose expansion, will receive the most appropriate dose and schedule identified from the first part of the study. More than one dose level or schedule from part 1 may be tested. Both the participants and the study team know what treatment the participants will take.

Participants in this study will take the study treatment 225Ac-pelgi once in a period of 6 weeks called a cycle. Each participant will have 4 of these treatment cycles, if the participant benefits from the treatment.

Each participant will be in the study for up to nearly six years, including a first test (screening) phase of a maximum of 30 days, up to 12 months of treatment depending on the participant's benefit, and a follow-up phase of 60 months after the end of treatment. The following visits to the study site are planned: 2 during the screening phase, 8 in the first treatment cycle, 7 in subsequent cycles, and a visit 6 to 12 weeks after the last dose. In the following 12 months, visits are planned every 6 weeks and during the next 48 months phone calls or clinic visits are planned approximately every 12 weeks.

In addition, a sub study during the dose escalation part will gather information on the distribution of the study treatment in the body, the proportion that binds to the cancer cells, and the resulting radiation at the tumor site.

During the study, the study team will:

* Do physical examinations
* Check vital signs such as blood pressure, heart rate, and body temperature
* Take blood, and urine samples
* Examine heart health using echocardiogram and electrocardiogram (ECG)
* Take tumor samples
* Track 225Ac-pelgi in the body using gamma imaging (generally available at all study sites)
* Check the tumor status using PET (positron emission tomography), CT (computed tomography) or MRI (magnetic resonance imaging) and bone scan
* Ask questions about the impact of the disease on the participants' wellbeing and activities of daily life (Eastern Cooperative Oncology Group Performance status (ECOG PS)).

ELIGIBILITY:
Inclusion Criteria:

* mCRPC with pathological confirmation of adenocarcinoma without small-cell or neuroendocrine features.
* Previous treatment with at least 1 Novel androgen axis drug (NAAD) (e.g., enzalutamide, apalutamide, darolutamide and/or abiraterone).
* Prior orchiectomy and/or ongoing androgen deprivation therapy and a castrate level of serum testosterone (<50 ng/dL or <1.7 nmol/L).
* Prior taxane treatment:

  * Dose Escalation: Participants must either have had prior treatment with at least 1 but no more than 2 taxane regimens, or been deemed ineligible for or refused taxane therapy on consultation with their physician
  * Dose Expansion Group A: Participants must have had prior treatment with at least 1 but no more than 2 taxane regimens, in the castration-resistant setting
  * Dose Expansion Group B: Participants must not have received taxane therapy since becoming castration-resistant
  * Dose Expansion Group C: Participants must either have had prior treatment with at least 1 but no more than 2 taxane regimens*, or been deemed ineligible for or refused taxane therapy on consultation with their physician *A taxane regimen consists of a minimum of 2 treatment cycles (maximum number of cycles as per local guidelines). A treatment break within a taxane regimen may be given provided that another anticancer therapy is not administered during that time
* Prior treatment with an established 177Lu-PSMA therapy (i.e., dose activity and cycles comparable to approved treatments) is required for participants in Dose Expansion Group C only. More specifically, to qualify for this expansion group, participants must not have discontinued 177Lu-PSMA tratment due to intolerance.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* Adequate bone marrow, hepatic, and renal function, as assessed by the following laboratory requirements within 30 days before start of study intervention:

  * Hemoglobin ≥9.0 g/dL
  * Absolute neutrophil count (ANC) ≥1500/mm^3
  * Platelet count ≥100,000/mm^3
  * Total bilirubin ≤1.5 x the Upper limit of normal (ULN), or <= 3 ULN if the participant has a confirmed history of Gilbert's syndrome (note that participants with Gilbert's syndrome should be carefully evaluated for other liver-related disorders that may impact their suitability for this study).
  * Alanine transaminase (ALT) and Aspartate transaminase (AST) ˂2.5 x ULN (≤5 x ULN for participants with liver involvement)
  * Participants on a stable dose of anticoagulation therapy are allowed to participate if they have no sign of bleeding or clotting, and Prothrombin time international normalized ratio (PT/INR) and activated partial thromboplastin time (aPTT) test results are acceptable at the Investigator's discretion
  * Estimated glomerular filtration rate (eGFR) >60 mL/min/1.73 m^2, according to the Modified Diet in Renal Disease (MDRD) abbreviated formula and creatinine clearance (CrCl) >60 mL/min based on Cockcroft-Gault formula
* Participants must have at least one Prostate-specific membrane antigen (PSMA)-positive distant metastatic lesion on the screening PSMA PET/CT scan using the study-designated PSMA PET tracers, as determined by the site Investigator. For eligibility purposes, a PSMA-positive lesion must have activity greater than the liver by visual assessment of the screening PSMA PET/CT. A PSMA-positive metastatic lesion should not correspond to a normal tissue structure or benign lesion.
* Documented progressive mCRPC per PCWG3, defined as meeting at least one of the following criteria:

  * PSA-progression (defined as 2 consecutive increases over a previous reference value obtained at a minimum of 1-week intervals, with a minimum starting value of 2.0 ng/mL)
  * Radiological progression in soft-tissue lesions according to PCWG3 modification of RECIST v1.1 criteria
  * Progression of bone disease (defined as ≥2 new bone lesions according to PCWG3 bone scan criteria).
  * Documented progressive mCRPC per PCWG3 and a minimun starting PSA value of 2.0 ng/mL is mandatory. Progressive mCRPC is defined as meeting at least one of the following criteria: a. PSA progression (defined as 2 consecutive increases over a previous reference value obtained at a minimun of 1-week intervals). b. Radiological progression in soft-tissue lesions according to PCWG3 modification of RECIST v1.1 criteria. c. Progression of bone disease (defined as ≥ 2 new bone lesions according to PCWG3 bone scan criteria).

Exclusion Criteria:

* Participants who have any of the following tumor lesions which are PSMA negative AND meet the size criteria below are excluded as determined by the site investigator. A PSMA-negative lesion for eligibility purposes must have activity equal to or less than the liver by visual assessment of the screening PSMA PET/CT scan using the study-designated PSMA PET/CT tracers. A PSMA-negative metastatic lesion should not correspond to a normal tissue structure or benign lesion.

  * a. Any single or multiple lymph node(s) ≥2.5cm in the short axis.
  * b. Any solid organ metastasis (e.g., lung, liver, adrenal glands, etc.) that is ≥1 cm in the short axis.
  * c. Any bone metastasis with a soft tissue component ≥ 1cm in short axis with the soft tissue component being PSMA-negative. PSMA-negative osseous metastases without a soft tissue component do not exclude a participant.
  * d. Predominantly necrotic lesions with greater than 1cm of enhancing tissue on contrast-enhanced Computer tomography / magnetic resonance imaging (CT/MRI).
* Prior systemic anticancer therapy including chemotherapy, NAAD, biologic therapy, immunotherapy, or investigational therapies within 4 weeks of the start of study intervention, except luteinizing hormone-releasing hormone (LHRH) or gonadotropin-releasing hormone (GnRH). Start of study intervention is allowed in shorter timeframes if 5 half-lives of the prior drug(s) have elapsed.
* Prior radiopharmaceutical treatment using actinium-225.
* Other prior radiopharmaceutical treatments:

  * Dose escalation and Dose expansion Groups A and B: Prior treatment with a radiopharmaceutical is prohibited.
  * Dose expansion Group C: Prior treatment with a radiopharmaceutical is prohibited with the following exceptions: Prior treatment with radium-223 dichloride more than 3 months before the start of study intervention is permitted; and prior treatment with 177Lu PSMA more than 6 weeks before the start of study intervention is required.

Note: Participants who have discontinued 177Lu-PSMA treatment due to intolerance are excluded from Group C.

* Prior definitive therapy (radiotherapy or surgery) completed less than 6 weeks before the start of study intervention. Note that palliative radiotherapy completed less than 6 weeks before the start of study intervention will be allowed if: (i) no more than 10% of the participants' bone marrow is irradiated, (ii) it does not encompass all potential target/measurable lesions for participants in dose expansion.
* Toxic effects of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥2 from prior anticancer therapy not yet stabilized or where significant post-treatment toxicities have been observed. Chronic toxic effects of CTCAE Grade ≤2 from prior anticancer therapy where no further resolution is expected do not require exclusion with agreement between the Investigator and Sponsor (e.g., chemotherapy-induced neuropathy, fatigue, alopecia, anorexia, etc.).
* Dose Expansion (Groups A, B and C): Presence of >3 liver metastases, any diffuse liver metastasis, or PSMA-non-avid liver metastasis (uptake is lower or equal compared to healthy liver tissue).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2031-08-10 (Estimated)

PRIMARY OUTCOMES:
Dose escalation & Dose expansion: The Incidence of treatment-emergent adverse events (TEAEs) including treatment-emergent serious adverse events (TESAEs) | After first administration of study treatment up to 42 days after the last dose of study treatment
Dose escalation & Dose expansion: The Severity of TEAEs including TESAEs | After first administration of study treatment up to 42 days after the last dose of study treatment
Dose escalation: Incidence of dose limiting toxicities (DLTs) at each 225Ac dose level during the DLT observation period | Up to Cycle 3 (each cycle is 42 days)
  DLTs will be summarized by MedDRA system organ class, preferred term and worst CTCAE grade.
Dose escalation: Objective response rate (ORR) at each 225Ac dose level during the DLT observation period | Up to Cycle 3 (each cycle is 42 days)
  ORR is defined as the proportion of participants who have a confirmed complete response (CR) or partial response (PR) per PCWG3 guidelines, as assessed by the Investigator.
Dose escalation: ≥50% decline in Prostate-specific antigen value from baseline (Cycle 1, Day 1) (PSA50) response at each 225Ac dose level during the DLT observation period | Up to Cycle 3 (each cycle is 42 days)
  PSA partial response is defined as a ≥50% decline in PSA value from Cycle 1 Day 1 (baseline). This PSA decline must be confirmed to be sustained by a second PSA value obtained 3 to 4 or more weeks later.
Dose expansion: Objective response rate (ORR) by Prostate Cancer Working Group 3 (PCWG3) guidelines based on investigator review | Up to 12 months after End of treatment
Dose expansion: ≥50% decline in Prostate-specific antigen value from baseline (Cycle 1, Day 1) (PSA50) response at 12 weeks or later | At 12 weeks or later (up to 12 months after End of treatment)
Dose expansion: Best overall Prostate-specific antigen (PSA) response | Up to 12 months after End of treatment

SECONDARY OUTCOMES:
Dose escalation & Dose expansion: Radiologic progression-free survival (rPFS ) by PCWG3 based on investigator review | Up to 12 months after end of treatment
  rPFS is defined as the time from the start of study treatment to the date of first observed disease progression (Investigator's radiological assessment by PCWG3) or death due to any cause, if death occurs before progression is documented.
Dose escalation & Dose expansion: Duration of PSA50 response | Up to 12 months after end of treatment
  Duration of PSA50 response by PCWG3 is defined as the time from the first documented PSA partial response as defined above to PSA progression by PCWG3 or death (if death occurs before progression is documented).
Dose escalation & Dose expansion: Duration of response (DOR) by PCWG3 based on investigator review | Up to 12 months after end of treatment
  DOR is defined as the time from the first documented objective response of PR or CR by PCWG3, whichever occurs earlier, to disease progression or death (if death occurs before progression is documented).
Dose escalation: Recommended dose level(s) of 225Ac-pelgi for dose expansion | Up to 4 cycles (each cycle is 42 days)
Dose escalation: Recommended dose schedule of 225Ac-pelgi for dose expansion | Up to 4 cycles (each cycle is 42 days)
Dose expansion: Recommended dose of 225Ac-pelgi for further clinical development | Up to 4 cycles (each cycle is 42 days)
Dose expansion: Recommended dose schedule of 225Ac-pelgi for further clinical development | Up to 4 cycles (each cycle is 42 days)
Dose escalation & Dose expansion: Maximum observed concentration (Cmax) of actinium-225 | Cycle 1, cycle 2 (From Pre-dose up to Day 36 post-dose for each cycle)
Dose escalation & Dose expansion: Maximum observed concentration (Cmax) of total antibody | Cycle 1, cycle 2 (From Pre-dose up to Day 36 post-dose for each cycle)
Dose escalation & Dose expansion: Area under the curve (AUC) of actinium-225 | Cycle 1, cycle 2 (From Pre-dose up to Day 36 post-dose for each cycle)
Dose escalation & Dose expansion: Area under the curve (AUC) of total antibody | Cycle 1, cycle 2 (From Pre-dose up to Day 36 post-dose for each cycle)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (5):
  - City of Hope - Duarte Cancer Center, Duarte, California
  - M Health Fairview Masonic Cancer Clinic - Clinics and Surgery Center, Minneapolis, Minnesota
  - XCancer Omaha, Omaha, Nebraska
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - Utah Cancer Specialists Cancer Center - Medical Oncology, Salt Lake City, Utah
- Canada (6):
  - Cross Cancer Institute, Clinical Trials Unit, Edmonton, Alberta
  - BC Cancer - Vancouver Site, Vancouver, British Columbia
  - Princess Margaret Cancer Centre - University Health Network - Department of Medical Oncology and Hematology, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre (MUHC) - Research Institute (RI) - McConnell Centre for Innovative Medicine (CIM), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke (CHUS) - Hopital Fleurimont, Sherbrooke, Quebec
- Finland (5):
  - Kuopio University Hospital, Kuopion yliopistollinen sairaala (KYS) - Syövänhoitokeskus, Kuopio, Northern Savonia
  - HUS-Yhtymä, Helsingin yliopistollinen sairaala (HUS) - Syöpäkeskus, Helsinki, Uusimaa
  - Docrates Mehiläinen Syöpäsairaala, Helsinki, Uusimaa
  - Tampere University Hospital, Tampereen yliopistollinen sairaala (TAYS) - Syöpäkeskus, Tampere
  - CRST Oy - Clinical Research Services Turku, Turku
- Italy (2):
  - Istituto Europeo di Oncologia s.r.l - Medicina Nucleare, Milan
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale - S. C. Medicina Nucleare e Terapia Metabolica, Napoli
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset - Klinisk prövningsenhet Fas I/FIH, Gothenburg
  - Skånes Universitetssjukhus Lund - Onkologens kliniska forskningsenhet, Lund
  - Karolinska Universitetssjukhuset - Fas I-enheten Solna CKC, Stockholm
  - Akademiska Sjukhuset - Fas-I-enheten, Uppsala
- Switzerland (3):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Univestitätsspital Zürich (USZ), Zurich
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust | Addenbrookes Hospital - Clinical Research Centre, Cambridge, Cambridgeshire
  - University College London Hospitals NHS Foundation Trust | University College Hospital - NIHR UCLH Clinical Research Facility, London, Greater London
  - The Royal Marsden NHS Foundation Trust | Sutton - Oak Foundation Drug Development Unit, Sutton, Surrey
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust | Freeman Hospital - Cancer Trials Research Centre, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Schatz CA, Zitzmann-Kolbe S, Moen I, Klotz M, Nair S, Stargard S, Bjerke RM, Wickstrom Biseth K, Feng YZ, Indrevoll B, Cruciani V, Karlsson J, Haendler B, Nielsen CH, Alfsen MZ, Hammer S, Hennekes H, Cuthbertson A, Hagemann UB, Larsen A. Preclinical Efficacy of a PSMA-Targeted Actinium-225 Conjugate (225Ac-Macropa-Pelgifatamab): A Targeted Alpha Therapy for Prostate Cancer. Clin Cancer Res. 2024 Jun 3;30(11):2531-2544. doi: 10.1158/1078-0432.CCR-23-3746. PMID 38593212
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/22143